CLINICAL TRIAL: NCT02331446
Title: Dose-response Effects of Different Volumes of Structured Exercise in the Inflammatory and Oxidative Stress Parameters in Postmenopausal Women: a Randomized Clinical Trial
Brief Title: The Effect of Different Volumes of Physical Exercise on the Immune System
Acronym: ProAFIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Matheus Pintanel Silva de Freitas, Masters course student, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 27371214.4.0000.5313
Record Dates: First submitted 2014-12-23; First posted 2015-01-06 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Immune System Diseases; Oxidative Stress
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): The control group will be oriented to maintain their normal activity and habits and will not receive the intervention.
- 90 minutes per week (Experimental): The group of 90 minutes per week will do three sessions of 30 minutes per week of concurrent training, which consists on 15 minutes of aerobic exercise and 15 minutes of strength training.
  Interventions: Behavioral: Physical exercise intervention
- 150 minutes per week (Experimental): The group of 150 minutes will do three sessions of 50 minutes per week, which consists on 25 minutes of aerobic exercise and 25 minutes of strength training.
  Interventions: Behavioral: Physical exercise intervention
- 210 minutes per week (Experimental): The group pf 210 minutes per week will do three sessions of 70 minutes per week, which consists on 35 minutes of aerobic exercise and 35 minutes of strength training.
  Interventions: Behavioral: Physical exercise intervention

INTERVENTIONS:
Behavioral: Physical exercise intervention
  Arms: 150 minutes per week; 210 minutes per week; 90 minutes per week

SUMMARY:
The investigators will do an intervention on four groups of previously sedentary post-menopausal women which consists: group 1 - 30 minutes per day of physical protocol; group 2 - 50 minutes per day of physical protocol; group 3 - 70 minutes per day of physical protocol; group 4 - sedentary control women. The protocol consists of three sessions per week of concurrent training (half session with aerobic training and the other part with weight training). Inflammatory and oxidative parameters will be analyzed and the investigators hypothesized that 90 minutes per week of concurrent training (group 1) will reduce the inflammatory parameters and the oxidative stress, and this improvements will be greater so much as the longer the sessions (a dose-response effect). The physical activity practiced out of the intervention will be controlled by a questionnaire (the commuting and leisure sections of the International Physical Activity Questionnaire) and the food intake by a 24-hour food recall.

DETAILED DESCRIPTION:
The protocol will consist of an intervention based on concurrent training, for previously sedentary post-menopausal women divided on four groups: 1) control group; 2) 90 minutes of physical training per week; 3) 150 minutes of training per week; 4) 210 minutes of training per week.

The control group will be oriented to maintain their normal activity and habits and will not receive the intervention. The group of 90 minutes per week will do three sessions of 30 minutes per week of concurrent training, which consists on 15 minutes of aerobic exercise and 15 minutes of strength training. The group of 150 minutes will do three sessions of 50 minutes per week, which consists on 25 minutes of aerobic exercise and 25 minutes of strength training. The group pf 210 minutes per week will do three sessions of 70 minutes per week, which consists on 35 minutes of aerobic exercise and 35 minutes of strength training.

The aerobic exercise will be performed on cycle-ergometers and the subjects will exercise between the levels 14 and 15 of Borg's scale of perceived exertion. The strength training will be performed on weight machines by a linear periodization, which will consist on a week of adaptation (series of 10 to 12 submaximal repetitions), next three weeks with series of 12 to 14 maximal repetitions, weeks five to eight with series of 10 to 12 maximal repetitions, weeks nine to twelve with series of eight to 10 maximal repetitions. Al participants will do the maximum number of series of strength training that the time permits.

The blood samples will be collected at the beginning of the study (week zero), at the middle (week six) and at the end (week 12). The subjects will fill a 24-hour food recall (to control the food intake) and the commuting and leisure sections of the International Physical Activity Questionnaire (to control the physical activity practiced out of the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Women have to be in the postmenopausal period, without physical disorders.

Exclusion Criteria:

* Women who answer positively to, at least, one of the issues of the PAR-Q instrument;
* Women with diabetes and/or cancer history;
* Women who underwent oophorectomy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matheus P Freitas, Principal Investigator — Federal University of Pelotas

RESULTS

PARTICIPANT FLOW:
Groups:
- 90 Minutes Per Week: The group of 90 minutes per week will do three sessions of 30 minutes per week of concurrent training, which consists on 15 minutes of aerobic exercise and 15 minutes of strength training.
  Physical exercise intervention
- 150 Minutes Per Week: The group of 150 minutes will do three sessions of 50 minutes per week, which consists on 25 minutes of aerobic exercise and 25 minutes of strength training.
  Physical exercise intervention
- 210 Minutes Per Week: The group pf 210 minutes per week will do three sessions of 70 minutes per week, which consists on 35 minutes of aerobic exercise and 35 minutes of strength training.
  Physical exercise intervention
Period: Overall Study
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Started | 9 | 11 | 11 | 11
Completed | 5 | 6 | 8 | 8
Not Completed | 4 | 5 | 3 | 3
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1
Not completed — Personal Problem | 2 | 0 | 0 | 0
Not completed — Disease | 0 | 2 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Lost before baseline analysis | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of baseline participants is not consistent with number provided in the Participant Flow module because two of the beginning participants did not arrived on the first data collection. Due to this, these participants (one of the 90 min/week, and other of the 150 min/week group) were lost to follow-up before the baseline data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week | Total
Number analyzed (Participants) | 9 | 10 | 10 | 11 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [63 to 73] | 62 [52 to 74] | 61.5 [59 to 67] | 63 [62 to 65] | 63 [60 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 11 | 40
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 3 | 9
  White | 7 | 8 | 8 | 8 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 9 | 10 | 10 | 11 | 40
Household Income [Median (Inter-Quartile Range); unit: US$] | 846 [612 to 1692] | 538 [338 to 846] | 867 [444 to 1269] | 423 [306 to 655] | 612 [338 to 1015]
Resting heart rate [Mean (Standard Deviation); unit: bpm] | 65.8 (7.9) | 64.7 (13.1) | 64.5 (9.2) | 68.1 (12.1) | 65.5 (10.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 119.8 (6.7) | 118.2 (20.4) | 121.2 (12.4) | 121.0 (14.2) | 120.8 (14.3)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.4 (8.8) | 75.2 (17.2) | 76.0 (7.0) | 78.7 (7.1) | 76.4 (10.6)
Marital status [Number; unit: participants]
  Married | 4 | 4 | 7 | 1 | 16
  Others | 5 | 6 | 3 | 10 | 24
Educational level [Number; unit: participants]
  Incomplete primary school | 1 | 4 | 3 | 4 | 12
  Primary school | 3 | 3 | 1 | 2 | 9
  Incomplete high school | 1 | 1 | 2 | 0 | 4
  High school | 3 | 1 | 4 | 2 | 10
  Incomplete higher education | 0 | 0 | 0 | 2 | 2
  Higher education | 1 | 1 | 0 | 1 | 3
Chronic Use of Medication [Number; unit: participants] — This variable refers to a chronic use of any medication.
  participants
    No | 0 | 1 | 1 | 1 | 3
    Yes | 9 | 9 | 9 | 10 | 37
Smoking [Number; unit: participants]
  No | 8 | 8 | 9 | 10 | 35
  Yes | 1 | 2 | 1 | 1 | 5
Alcohol intake [Number; unit: participants]
  Daily (one dose) | 0 | 0 | 1 | 0 | 1
  Sporadically | 5 | 4 | 7 | 5 | 21
  No | 4 | 6 | 2 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin-6
Time Frame: Weeks 0, 6 and 12
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
pg/mL
  Baseline | 4.60 [3.96 to 5.77] | 4.58 [3.62 to 4.88] | 4.50 [3.84 to 6.35] | 5.27 [4.05 to 13.01]
  Week 6 | 3.62 [3.42 to 4.41] | 4.14 [3.54 to 4.29] | 4.39 [4.06 to 4.87] | 4.67 [3.67 to 6.69]
  Week 12 | 4.47 [4.26 to 4.54] | 3.82 [3.57 to 8.92] | 4.71 [3.46 to 5.39] | 5.55 [3.97 to 7.01]

2. Primary Outcome: Change in Adenosine Deaminase Activity
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
U/L
  Baseline | 31.12 (5.96) | 29.94 (11.72) | 31.83 (5.84) | 25.91 (8.45)
  Week 6 | 42.11 (10.74) | 42.54 (10.07) | 42.34 (11.53) | 45.03 (9.05)
  Week 12 | 43.11 (20.21) | 45.89 (9.75) | 37.83 (10.51) | 47.70 (17.90)

3. Primary Outcome: Change in Butyrylcholinesterase Activity
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: µmol BuSCh/h/mg of protein
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
µmol BuSCh/h/mg of protein
  Baseline | 9.35 (2.79) | 10.83 (2.00) | 7.44 (4.31) | 7.31 (4.23)
  Week 6 | 10.07 (0.83) | 11.46 (2.83) | 9.40 (2.85) | 11.02 (2.83)
  Week 12 | 11.16 (1.65) | 9.49 (1.28) | 8.71 (1.78) | 10.34 (2.77)

4. Primary Outcome: Change in Thiobarbituric Acid Reactive Substances
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: nmol TBARS/mg protein
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
nmol TBARS/mg protein
  Baseline | 0.100 (0.022) | 0.144 (0.039) | 0.131 (0.028) | 0.137 (0.017)
  Week 6 | 0.119 (0.020) | 0.159 (0.053) | 0.162 (0.049) | 0.149 (0.018)
  Week 12 | 0.073 (0.040) | 0.095 (0.020) | 0.062 (0.024) | 0.070 (0.019)

5. Primary Outcome: Change in Total Thiol Content
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: nmol TNB/mg protein
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
nmol TNB/mg protein
  Baseline | 9.00 (1.45) | 7.74 (0.94) | 7.73 (1.85) | 7.07 (1.63)
  Week 6 | 12.26 (2.50) | 12.10 (3.69) | 12.42 (4.31) | 12.13 (3.65)
  Week 12 | 9.24 (1.44) | 8.55 (2.53) | 7.80 (1.51) | 8.32 (1.52)

6. Primary Outcome: Change in Glutathione Peroxidase Activity
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: U/mg protein
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
U/mg protein
  Baseline | 87.32 (15.68) | 63.69 (41.12) | 73.53 (40.56) | 65.31 (29.52)
  Week 6 | 90.24 (11.99) | 91.26 (44.79) | 80.57 (43.76) | 98.87 (33.17)
  Week 12 | 93.08 (13.84) | 81.72 (12.52) | 80.04 (18.26) | 77.32 (13.01)

7. Secondary Outcome: Change in Performance in the Six-minute Walk Test
Time Frame: Weeks 0 and 12
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
Meters
  Baseline | 466.49 (97.89) | 515.78 (69.08) | 552.62 (62.29) | 539.77 (46.17)
  Week 12 | 514.5 (124.24) | 581.02 (76.02) | 559.57 (53.03) | 586.69 (66.53)

8. Secondary Outcome: Change in Handgrip Strength
Description: Measured using a handgrip dynamometer and quantified in kilogram-force
Time Frame: Weeks 0 and 12
Measure: Mean (Standard Deviation); unit: kgf
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
kgf
  Baseline | 23.61 (3.91) | 23.80 (5.46) | 25.03 (5.70) | 24.81 (4.23)
  Week 12 | 22.98 (4.92) | 26.56 (5.76) | 26.67 (6.64) | 30.39 (4.19)

9. Other Pre Specified Outcome: Change in Body Mass Index
Time Frame: Weeks 0 and 12
Measure: Median (Inter-Quartile Range); unit: kg/m²
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
kg/m²
  Baseline | 29.69 [28.14 to 34.98] | 28.25 [23.84 to 31.96] | 28.62 [23.61 to 30.44] | 29.56 [24.49 to 30.68]
  Week 12 | 28.09 [27.35 to 31.12] | 28.03 [23.71 to 29.61] | 28.97 [24.54 to 30.15] | 28.20 [24.74 to 32.4]

10. Other Pre Specified Outcome: Change in Minutes Per Week of Physical Activity Out of Intervention
Description: Measured by the commuting and leisure sections of the International Physical Activity Questionnaire
Time Frame: Week 0 and 12
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
minutes per week
  Baseline | 30 [0 to 120] | 35 [0 to 200] | 60 [0 to 120] | 150 [80 to 300]
  Week 12 | 90 [40 to 120] | 90 [60 to 90] | 65 [20 to 125] | 150 [60 to 240]

11. Other Pre Specified Outcome: Change in Calories Intake
Description: Measured by a 24-hour food recall and quantified in calories
Time Frame: Weeks 0 and 12
Measure: Mean (Standard Deviation); unit: cal
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
cal
  Baseline | 1700.45 (178.56) | 1390.64 (687.00) | 1461.53 (544.92) | 1485.54 (474.46)
  Week 12 | 1873.03 (531.22) | 1720.32 (534.82) | 1229.61 (550.19) | 1322.39 (317.85)

12. Other Pre Specified Outcome: Educational Level
Description: Measured by a questionnaire and quantified categorically in: Incomplete primary school; Primary school; Incomplete high school; High school; Incomplete higher education; Higher education. The number of baseline participants is not consistent with number provided in the Participant Flow module because two of the beginning participants did not arrived on the first data collection. Due to this, these participants (one of the 90 min/week, and other of the 150 min/week group) were lost to follow-up before the baseline data collection.
Time Frame: Week 0
Measure: Number; unit: participants
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 9 | 10 | 10 | 11
participants
  Incomplete primary school | 1 | 4 | 3 | 4
  Primary school | 3 | 3 | 1 | 2
  Incomplete high school | 1 | 1 | 2 | 0
  High school | 3 | 1 | 4 | 2
  Incomplete higher education | 0 | 0 | 0 | 2
  Higher education | 1 | 1 | 0 | 1

13. Other Pre Specified Outcome: Household Income
Description: Measured by a questionnaire and quantified by the income of all persons in the participant's home. The number of baseline participants is not consistent with number provided in the Participant Flow module because two of the beginning participants did not arrived on the first data collection. Due to this, these participants (one of the 90 min/week, and other of the 150 min/week group) were lost to follow-up before the baseline data collection.
Time Frame: Week 0
Measure: Median (Inter-Quartile Range); unit: US$
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 9 | 10 | 10 | 11
US$ | 846 [612 to 1692] | 538 [338 to 846] | 867 [444 to 1269] | 423 [306 to 655]

14. Other Pre Specified Outcome: Age
Description: The number of baseline participants is not consistent with number provided in the Participant Flow module because two of the beginning participants did not arrived on the first data collection. Due to this, these participants (one of the 90 min/week, and other of the 150 min/week group) were lost to follow-up before the baseline data collection.
Time Frame: Week 0
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 9 | 10 | 10 | 11
years | 70 [63 to 73] | 62 [52 to 74] | 61.5 [59 to 67] | 63 [62 to 65]

15. Other Pre Specified Outcome: Chronic Use of Medication
Description: Measured by a questionnaire and quantified categorically in: No; Yes. This variable refers to a chronic use of any medication. The number of baseline participants is not consistent with number provided in the Participant Flow module because two of the beginning participants did not arrived on the first data collection. Due to this, these participants (one of the 90 min/week, and other of the 150 min/week group) were lost to follow-up before the baseline data collection.
Time Frame: Week 0
Measure: Number; unit: participants
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 9 | 10 | 10 | 11
participants
  No | 0 | 1 | 1 | 1
  Yes | 9 | 9 | 9 | 10

16. Primary Outcome: Change in Superoxide Dismutase Activity
Time Frame: Weeks 0, 6 and 12
Measure: Mean (Standard Deviation); unit: U/mg protein
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Number analyzed (Participants) | 5 | 6 | 8 | 8
U/mg protein
  Baseline | 6.10 (1.33) | 5.31 (0.79) | 5.72 (1.44) | 4.67 (1.11)
  Week 6 | 6.04 (0.62) | 5.04 (1.67) | 4.20 (0.79) | 5.02 (1.15)
  Week 12 | 6.36 (0.31) | 4.79 (1.29) | 4.86 (1.06) | 4.78 (1.46)

ADVERSE EVENTS:
Arm/Group | Control | 90 Minutes Per Week | 150 Minutes Per Week | 210 Minutes Per Week
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
The test performed to estimate the cardiorespiratory fitness was not specific to measure physical activity performed by the women. The test was done walking (six-minute walking test) and the aerobic training was carried out on cycle-ergometers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No